CLINICAL TRIAL: NCT04178980
Title: Double-blinded, Randomized Controlled Trial of Simvastatin Use As Adjuvant Therapy in Relapsing-Remitting Multiple Sclerosis
Brief Title: Role of Simvastatin in Relapsing-Remitting Multiple Sclerosis
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mena Mahfouz Fahim, researcher, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: simvastatin in MS
Record Dates: First submitted 2019-11-25; First posted 2019-11-26 (Actual); Last update posted 2019-11-29 (Actual); Status verified 2019-11

CONDITIONS: Simvastatin Multiple Sclerosis
MeSH Terms: interventions — Simvastatin

STUDY DESIGN:
Intervention Model Description: double blinded
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- case (Active Comparator)
  Interventions: Drug: Simvastatin in relapsing remitting multiple sclerosis
- control (Placebo Comparator)
  Interventions: Drug: Simvastatin in relapsing remitting multiple sclerosis

INTERVENTIONS:
Drug: Simvastatin in relapsing remitting multiple sclerosis — Simvastatin use as adjuvant thearapy in relapsing remitting multiple sclerosis

SUMMARY:
The purpose of the clinical trial is to test how Simvastatin (80mg/day) may decrease attacks and progression of disease in patients with multiple sclerosis under disease modifying therapy (DMTs)

DETAILED DESCRIPTION:
Multiple sclerosis (MS), the most prevalent neurological disability, is an autoimmune-mediated disorder that affects the central nervous system (CNS) and often leads to severe physical or cognitive incapacitation as well as neurological problems in young adults . Multifocal zones of inflammation due to focal T-lymphocytic and macrophage infiltrations, and oligodendrocyte death are the primary causes of myelin sheath destruction (2) that result in the formation of CNS plaques composed of inflammatory cells and their products, demyelinated and transected axons, and astrogliosis in both white and gray matter. These lesions can cross-talk with the correct transmission of nerve impulses and lead to neuronal dysfunction such as autonomic and sensorimotor defects, visual disturbances, ataxia, fatigue, difficulties in thinking, and emotional problems .

Subtypes of MS are considered important not only for prognosis but also for treatment decisions and include:

* Relapsing remitting MS (RRMS)
* Primary progressive MS (PPMS)
* Secondary progressive MS (SPMS)
* Progressive relapsing MS (PRMS). RRMS is the most common subtype (approximately 87%) which characterized by unpredictable acute attacks followed by periods of remission . During RRMS, inflammatory attacks on myelin and nerve fibers occur. Activated immune cells cause lesions in the CNS which generate symptoms of visual impairments, tingling and numbness, episodic bouts of fatigue, intestinal and urinary system disorders, spasticity, and learning and memory impairment. Approximately 10-15% of MS patients are diagnosed with PPMS which largely affect the nerves of the spinal cord. PPMS patients tend to have fewer brain lesions. Induced symptoms include problems with walking, weakness, stiffness, and trouble with balance.

Nearly 65% of patients with RRMS will subsequently develop SPMS which is considered the second phase of this disease. Many individuals experience increased weakness, intestinal and urinary system disorders, fatigue, stiffness, mental disorders, and psychological impairment. Finally, PRMS is the least common type of MS that occurs in approximately 5% of patients and is associated with symptoms such as eye pain and double vision, along with sexual, intestinal and urinary system dysfunction, dizziness, and depression. Generally MS is detected between the ages of 20 and 40 years, but less than 1% can occur in childhood and approximately 2-10% after 50 years of age .

This pathologic condition affects women more than men (sex ratio 2.5:1) and the prevalence varies by geographic area, ranging from 120 per 100,000 individuals . The etiology of MS remains unclear, however it can be considered a multifactorial disease and include a genetic predisposition combined with environmental influences .

The initial treatment strategy for MS is largely based on disease-modifying drugs such as interferon-β and glatiramer acetate . The effects of these treatments are partially for symptomatic alleviation and do not stop the ongoing neurodegeneration.

Simvastatin Simvastatin belongs to a group of medicines called statins. Its action is inhibiting 3-hydroxy-3-methylglutaryl (HMG) coenzyme A reductase. HMG-CoA reductase, the rate-limiting enzyme of the HMG-CoA reductase pathway, the metabolic pathway responsible for the endogenous production of cholesterol. Statins are more effective than other lipid-regulating drugs at lowering LDL-cholesterol concentration Furthermore, simvastatin has pleiotropic effects associated with onset and progression of autoimmune and inflammatory diseases, cancer, neurodegenerative disorders, strokes, bacterial infections, and human immunodeficiency virus. Understanding these issues will improve the prognosis of patients who are administered statins and potentially expand our ability to treat a wide variety of diseases .

Simvastatin was found to decrease the incidence of hemodynamically significant rejection episodes in cardiac transplant patients. This effect was not significantly correlated to reduction in cholesterol levels in these patients. Subsequent studies have revealed many immunological pathways sensitive to modulation by statins:

1. Simvastatin inhibit interferon-γ-inducible class II transactivator (CIITA) to decrease the induction/up regulation of MHC class II molecules on professional & non- professional antigen presenting cells.
2. Statins bind to β2 integrin and thereby block T-cell co-stimulation by means of lymphocyte function-associated antigen-1 (LFA-1).
3. In monocytes and macrophages, statins decrease chemotaxis, lipopolysaccharide (LPS) mediated release of tumour necrosis factor-α (TNF-α), activation of NO synthase8 and LPS-stimulated secretion of matrix metalloproteinase-9 (12).

Common simvastatin side effects may include:

* Headache;
* Constipation, nausea, stomach pain; or
* Cold symptoms such as stuffy nose, sneezing, sore throat.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients must have a confirmed diagnosis of multiple sclerosis according to revised Mc Donald criteria 2017 and have relapsing remitting multiple scelerosis type.

  2. EDSS up to 4. 3. Males and Females aged 18 to 65 4. pregnancy test within 7 days prior to being registered/randomized. Participants are considered not of child bearing potential if they are surgically sterile (i.e. they have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are postmenopausal.

  5. Willing and able to comply with the trial protocol (e.g. can tolerate MRI and fullfills the requirements for MRI, e.g. not fitted with pacemakers or permanent hearing aids), with ability to understand and complete questionnaires 6. Willing and able to provide written informed consent

Exclusion Criteria:

* 1. Unable to give informed consent. 2. Patient with other types of multiple scelerosis (Secondary-Progressive MS (SPMS), Primary progressive MS, Progressive-Relapsing MS (PRMS) ) 3. Any medications that unfavourably interact with statins e.g.: fibrates, nicotinic acid, cyclosporin, azole anti-fungal preparations, macrolideantibiotics, protease inhibitors, nefazodone, verapamil, amiodarone, large amounts of grapefruit juice or alcohol abuse within 6 months.

  4. Active Hepatic disease or known severe renal failure (creatinine clearance <30ml/min) 5. Screening levels of alanine aminotransferase (ALT), aspartate aminotransferase (AST) or creatine kinase (CK) are three times the upper limit of normal patients.

  6. Patient unable to tolerate or unsuitable to have baseline MRI scan (e.g. metal implants, heart pacemaker) or MRI scan not of adequate quality for analysis (e.g. too much movement artefact).

  7. Females who are pregnant, planning pregnancy or breastfeeding. 8. Allergy to simvastatin

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
EDSS | baseline, month 6, 12, 18, 24
  Time to confirmed disability progression between simvastatin and placebo arm based on change in EDSS scores compared to baseline

SECONDARY OUTCOMES:
Response rate on the patient reported outcome form Multiple Sclerosis Walking Scale-12 version 2 | baseline, month 12 and 24
  MSWS-12v2 is a12 item patient report measure on the impact of MS on the individual's walking ability over the previous 2 weeks. Each item will be summed to generate a total score and transformed to a scale with a range of 0 to 100 with high scores indicating greater impact on walking.
Change in time taken to complete 25-Foot Timed Walk | baseline, month 6, 12, 18 and 24
  a quantitative mobility and leg function performance test based on a timed 25-foot walk
Change in time taken to complete 9 hole peg test | baseline, month 6, 12, 18 and 24
  a brief, standardized, quantitative test of upper extremity function. Participants are instructed to pick up 9 pegs, one at a time, as quickly as possible and are required to insert them into 9 empty peg holes. Once all nine pegs have been inserted, the participant should immediately remove the pegs, one at a time. The total time taken to complete the task is recorded. Two consecutive trials with the dominant hand are immediately followed by two consecutive trials with the non-dominant hand. The two trials for each hand are averaged.
modified Rankin scale | baseline, month 12 and 24
  is used to evaluate the degree of disability in daily activities of those with neurological disability
Change in frontal lobe function based on Frontal Assessment Battery (FAB) scores | baseline, month 12 and 24
  brief battery of six neuropsychological tasks designed to assess frontal lobe function. The six FAB tasks assess conceptualisation (abstract reasoning), item flexibility (verbal fluency), motor programming (organisation, maintenance and execution of successive actions), sensitivity to interference (conflicting instructions), inhibitory control (inhibit inappropriate responses), and environmental autonomy. The test takes approximately 10 minutes to complete.

REFERENCES:
- [Background] Loma I, Heyman R. Multiple sclerosis: pathogenesis and treatment. Curr Neuropharmacol. 2011 Sep;9(3):409-16. doi: 10.2174/157015911796557911. PMID 22379455
- [Background] Gadoth N. Multiple sclerosis in children. Brain Dev. 2003 Jun;25(4):229-32. doi: 10.1016/s0387-7604(03)00035-4. PMID 12767451
- [Background] Boiko A, Vorobeychik G, Paty D, Devonshire V, Sadovnick D; University of British Columbia MS Clinic Neurologists. Early onset multiple sclerosis: a longitudinal study. Neurology. 2002 Oct 8;59(7):1006-10. doi: 10.1212/wnl.59.7.1006. PMID 12370453
- [Background] Haas J, Korporal M, Balint B, Fritzsching B, Schwarz A, Wildemann B. Glatiramer acetate improves regulatory T-cell function by expansion of naive CD4(+)CD25(+)FOXP3(+)CD31(+) T-cells in patients with multiple sclerosis. J Neuroimmunol. 2009 Nov 30;216(1-2):113-7. doi: 10.1016/j.jneuroim.2009.06.011. Epub 2009 Jul 31. PMID 19646767
- [Background] Fisk JD, Ritvo PG, Ross L, Haase DA, Marrie TJ, Schlech WF. Measuring the functional impact of fatigue: initial validation of the fatigue impact scale. Clin Infect Dis. 1994 Jan;18 Suppl 1:S79-83. doi: 10.1093/clinids/18.supplement_1.s79. PMID 8148458